CLINICAL TRIAL: NCT00958880
Title: Placebo-Controlled Evaluation of the Efficacy of Yohimbine Hydrochloride for Enhancing the Effects of CBT for Social Phobia
Brief Title: Yohimbine to Enhance Cognitive Behavioral Therapy (CBT) for Social Anxiety
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Southern Methodist University (Other)
Responsible Party: Principal Investigator, Jasper Smits, Ph.D., Principal Investigator, Southern Methodist University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KS09-088; KS09-088
Record Dates: First submitted 2009-08-12; First posted 2009-08-13 (Estimated); Results first posted 2013-11-11 (Estimated); Last update posted 2013-11-11 (Estimated); Status verified 2013-09

CONDITIONS: Social Anxiety Disorder
MeSH Terms: conditions — Phobia, Social | interventions — Yohimbine; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sugar Pill (Placebo Comparator): Participants will receive placebo (sugar pill) augmented Group Cognitive Behavioral Therapy
  Interventions: Behavioral: Group Cognitive Behavioral Therapy; Drug: Sugar Pill
- Yohimbine Hydrochloride (Experimental): Participants will receive Yohimbine Hydrochloride augmented Group Cognitive Behavioral Therapy
  Interventions: Behavioral: Group Cognitive Behavioral Therapy; Drug: Yohimbine Hydrochloride

INTERVENTIONS:
Behavioral: Group Cognitive Behavioral Therapy — 5 weeks of group CBT for Social Anxiety. The aim of CBT is to help participants become more comfortable with social situations
  One arm will receive placebo augmented Group Cognitive Behavioral Therapy and the other will receive yohimbine hydrochloride augmented cognitive behavioral therapy.
Drug: Yohimbine Hydrochloride — Participants in the Yohimbine augmented arm will receive 4 doses of Yohimbine Hydrochloride before 4 of the 5 group cognitive behavioral therapy sessions.
  Arms: Yohimbine Hydrochloride
Drug: Sugar Pill — Participants in the placebo (sugar pill) augmented arm will receive 4 doses of a sugar pill before 4 of the 5 group cognitive behavioral therapy sessions.
  Arms: Sugar Pill

SUMMARY:
The purpose of this study is to investigate the utility of Yohimbine hydrochloride for facilitating fear extinction in a sample of patients with social phobia who will be treated with CBT.

DETAILED DESCRIPTION:
The primary aim is to determine the relative efficacy of exposure-based CBT for social phobia when conducted with adjunctive acute (prior to four of five sessions) administration of either Yohimbine hydrochloride (10.8 mg) or placebo during core exposure sessions. Based on the available evidence, the investigators hypothesize that acute treatment with Yohimbine hydrochloride prior to exposure-based CBT would facilitate the extinction of fear that occurs with this treatment and would enhance treatment outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female outpatients between 18 and 65 years of age with a primary psychiatric diagnosis (designated by the patient as the most important source of current distress) of non-generalized social anxiety disorder (SAD) or Generalized Social Anxiety Disorder (GSAD) with a significant fear of public speaking as defined by DSM-IV criteria.
2. Severity of the social phobia of at least 3 on the CGI scale rated for the severity of public speaking anxiety
3. Willingness and ability to comply with the requirements of the study protocol.

Exclusion Criteria:

1. A lifetime history of bipolar disorder, schizophrenia, psychosis, delusional disorders or obsessive-compulsive disorder; an eating disorder in the past 6 months; organic brain syndrome, mental retardation or other cognitive dysfunction that could interfere with capacity to engage in therapy; a history of substance (amphetamines, benzodiazepines, barbiturates, cocaine metabolites, marijuana, narcotics, and sedative hypnotics) abuse or dependence or alcohol abuse or dependence (other than nicotine) in the last 6 months or otherwise unable to commit to refraining from alcohol use during the acute period of study participation.
2. Patients with posttraumatic stress disorder within the past 6 months are excluded. Entry of patients with other mood or anxiety disorders will be permitted if the social anxiety disorder is judged to be the predominant disorder, in order to increase accrual of a clinically relevant sample. Patients with significant suicidal ideation (BDI item 9 score > 1) or who have enacted suicidal behaviors within 6 months prior to intake will be excluded from study participation and referred for appropriate clinical intervention.
3. Given that Yohimbine hydrochloride is frequently used as an adjunctive medication in order to decrease side effects commonly resulting from antidepressant use (Pollack & Smoller, 1996), antidepressant and anxiolytic medications are acceptable if they are stabilized for at least 8 weeks prior to the baseline assessments. However, individuals taking monoamine oxidase inhibitors or tricyclic antidepressants will be excluded from the study unless they are able and willing to discontinue these medications prior to baseline screening.
4. Individuals taking antihistamines or strattera (atomoxetine) will be excluded from the study unless they are able and willing to discontinue these medications prior to baseline screening
5. Evidence through interview or physical exam of significant general medical condition (e.g renal, endocrine, hepatic, respiratory, cardiovascular, hematologic, immunologic or cerebrovascular disease, or malignancy) that may interfere with the interpretation of safety and efficacy evaluations in the opinion of the prescribing physician.
6. Resting blood pressure ≥ 160 systolic and/or 100 diastolic. Individuals currently being treated for high blood pressure and meeting these criteria are eligible.
7. Significant personality dysfunction likely to interfere with study participation.
8. Patients with a current or past history of seizures
9. Pregnant women, lactating women, and women of childbearing potential who are not using medically accepted forms of contraception (e.g., IUD, oral contraceptives, barrier devices, condoms and foam, or implanted progesterone rods stabilized for at least 3 months). A urine pregnancy test will be performed on all female subjects of child-bearing potential at the screening visit.
10. Any concurrent psychotherapy initiated within 3 months of baseline, or ongoing psychotherapy of any duration directed specifically toward treatment of the SAD is excluded. Prohibited psychotherapy includes CBT or psychodynamic therapy focusing on exploring specific, dynamic causes of the phobic symptomatology and provides management skills. General supportive therapy initiated > 3 months prior is acceptable.
11. Prior non-response to adequately-delivered exposure (i.e., as defined by the patient's report of receiving specific and regular exposure assignments as part of a previous treatment) will exclude participants from the study.
12. Patients with a history of head trauma causing loss of consciousness, seizure or ongoing cognitive impairment.
13. Patients unable to understand study procedures and participate in the informed consent process.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-03; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jasper Smits, Ph.D., Principal Investigator — Southern Methodist University; Michael W Otto, Ph.D., Principal Investigator — Boston University
Locations (2):
- United States (2):
  - Boston University, Boston, Massachusetts
  - Southern Methodist University, Dallas, Texas

REFERENCES:
- [Background] Powers MB, Smits JA, Otto MW, Sanders C, Emmelkamp PM. Facilitation of fear extinction in phobic participants with a novel cognitive enhancer: a randomized placebo controlled trial of yohimbine augmentation. J Anxiety Disord. 2009 Apr;23(3):350-6. doi: 10.1016/j.janxdis.2009.01.001. Epub 2009 Jan 15. PMID 19223151
- [Derived] Smits JA, Rosenfield D, Davis ML, Julian K, Handelsman PR, Otto MW, Tuerk P, Shiekh M, Rosenfield B, Hofmann SG, Powers MB. Yohimbine enhancement of exposure therapy for social anxiety disorder: a randomized controlled trial. Biol Psychiatry. 2014 Jun 1;75(11):840-6. doi: 10.1016/j.biopsych.2013.10.008. Epub 2013 Oct 16. PMID 24237691
- See also: BU Center for Anxiety and Related Disorders — http://www.bu.edu/anxiety

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were screened for eligibility criteria using an online screen. Potentially eligible participants were invited to the laboratory for a psychiatric interview. Eligible participants were enrolled in the Dallas area from 2009 to 2012.
Pre-assignment Details: Participants were not enrolled if they did not meet the study inclusion criteria at a psychiatric screening or medical evaluation designed to rule out contraindicated psychiatric or medical conditions.
Groups:
- Sugar Pill: Participants received placebo (sugar pill) augmented Group Cognitive Behavioral Therapy. The pills were administered 1 hour prior to sessions 2-5 of a 5-session group exposure-based CBT protocol.
- Yohimbine Hydrochloride: Participants received Yohimbine Hydrochloride augmented Group Cognitive Behavioral Therapy. Participants received Yohimbine HCL augmented Group Cognitive Behavioral Therapy. The 10.8 mg pills were administered 1 hour prior to sessions 2-5 of a 5-session group exposure-based CBT protocol.
Period: Overall Study
Arm/Group | Sugar Pill | Yohimbine Hydrochloride
Started | 20 | 20
Completed | 18 | 18
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sugar Pill | Yohimbine Hydrochloride | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 40
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 38.70 (12.08) | 35.50 (14.02) | 36.13 (12.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 5 | 14
  Male | 11 | 15 | 26
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: The Liebowitz Social Anxiety Scale (LSAS)
Description: The Liebowitz Social Anxiety Scale (LSAS) is a self-report measure of social anxiety symptom severity. Scores range from 0 to 144, with higher scores indicating more social anxiety symptoms severity (i.e., a worse outcome).
Time Frame: LSAS means at 1 month follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sugar Pill | Yohimbine Hydrochloride
Number analyzed (Participants) | 20 | 20
units on a scale | 41.0 (22.0) | 33.3 (17.5)
Statistical Analysis 1: Comparison: Sugar Pill vs Yohimbine Hydrochloride; Test type: Superiority or Other; p = .015, Regression, Linear; Slope = 10.46

2. Secondary Outcome: Social Phobic Disorders Severity and Change Form
Description: Social Phobic Disorders Severity and Change (SPDSC) Form is a version of the Clinical Global Improvement-Severity scale adapted specifically for clinician ratings of social anxiety disorder symptom severity. The scale ranges from 0 to 5, with higher scores indicating more social anxiety symptoms severity (i.e., worse outcomes). We examined the change in SPDSC scores from baseline to a 1 month follow-up.
Time Frame: CGI change scores from baseline to 1 month follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sugar Pill | Yohimbine Hydrochloride
Number analyzed (Participants) | 20 | 20
units on a scale | 2.0 (0.9) | 2.0 (0.8)
Statistical Analysis 1: Comparison: Sugar Pill vs Yohimbine Hydrochloride; Test type: Superiority or Other; p = .575, Regression, Linear; Slope = .03

ADVERSE EVENTS:
Arm/Group | Sugar Pill | Yohimbine Hydrochloride
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 5/20 | 19/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sugar Pill (N=20) | Yohimbine Hydrochloride (N=20)
Sweaty palms (General disorders) | 1 (1) | 0 (0)
Headache (General disorders) | 3 (3) | 2 (2)
Decrease in sexual arousal (General disorders) | 1 (1) | 0 (0)
Insomnia (General disorders) | 0 (0) | 2 (2)
Crying (General disorders) | 0 (0) | 1 (1)
Jittery/Jumpy (General disorders) | 0 (0) | 2 (2)
Tiredness (General disorders) | 0 (0) | 1 (1)
Light-headedness (General disorders) | 0 (0) | 1 (1)
Sweating (General disorders) | 0 (0) | 1 (1)
Alertness (General disorders) | 0 (0) | 1 (1)
Dazed (General disorders) | 0 (0) | 1 (1)
Heart palpitations (General disorders) | 0 (0) | 1 (1)
Hunger (General disorders) | 0 (0) | 1 (1)
Anxiety (General disorders) | 0 (0) | 2 (2)
Open sinuses (General disorders) | 0 (0) | 1 (1)
Hot flash/chills (General disorders) | 0 (0) | 6 (6)
Nausea (General disorders) | 0 (0) | 3 (3)
Pressure around the eyes (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No